CLINICAL TRIAL: NCT02649907
Title: Analysis of the Variability of Appetite and Energy Regulating Hormones to an Acute Nutritive Stimulation by Different Combinations of Macronutrients
Brief Title: Effects of Weight Loss on Nutritional Mediated Hormone Secretion
Acronym: RepDiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Knut Mai, Prof. Dr. med. Knut Mai (Principal Investigator and Clinical Professor, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA1/143/15
Record Dates: First submitted 2015-11-04; First posted 2016-01-08 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Weight Loss; Hormone Disturbance; Weight Gain
MeSH Terms: conditions — Weight Loss; Endocrine System Diseases; Weight Gain | interventions — Nutrition Assessment; Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Weight loss (Experimental): 3 months weight loss intervention by behavioral intervention
  Interventions: Dietary Supplement: nutritional stimulation via different testmeals; Other: Nutritional counseling; Dietary Supplement: formula diet

INTERVENTIONS:
Dietary Supplement: nutritional stimulation via different testmeals — nutritional stimulation of hormonal response through different testmeals
Other: Nutritional counseling — nutritional counseling for healthy eating behaviour
Dietary Supplement: formula diet — formula diet to help weight loss

SUMMARY:
Investigative trial with aim of

1. the description of the hormonal and metabolic response to meals containing different compositions of macronutrients
2. the metabolic response to these test meals in dependance of the hepatic and muscular insulin sensitivity and abdominal adipose tissue and
3. effects of a weight loss on the hormonal response to these test meals containing different compositions of macronutrients

Primary endpoint:

Glucagon-like-peptide 1 (GLP-1), Glucose dependent insulinotropic peptide (GIP) and Ghrelin response to a nutritive stimulation characterized by different nutritional composition

Secondary endpoints:

* differences of substrate utilization depending on the nutritive composition
* effects of different hepatic and muscular insulin sensitivity as well as impact of visceral fat mass on the hormonal and metabolic response
* effect of weight loss on the hormonal and metabolic response to different test meals

Study procedure:

After primary characterization 50 probands (male and female) will receive 3 different test meals within a randomised (meal order) controlled trial.

The three different test meals differ in nutritional composition. During consumption of the test meal a characterization of the endogenous hormonal response and appetite behaviour is performed.

A nutritional counselling is performed according to the guidelines of the German Nutrition Society (DGE) to ensure a stable nutritive behaviour in the three days before the test meal administration.

After analysis of the hormonal response to these 3 different testmeals follows a weight reduction period over 3 months. Afterwards reevaluation of the probands (again administration of 3 different test meals over a period of 3 weeks) will be performed.

Principal aim of the study:

Gain of information leading to the understanding of the hormonal regulation of food intake. The individual variability shall be determined with the aim of an identification of patient groups which show various intensities of the responses to different macronutrients.

ELIGIBILITY:
Inclusion Criteria:

* BMI>27 kg/m2
* given written informed consent

Exclusion Criteria:

* type 2 diabetes patients treated by insulin or drugs influencing incretin levels
* lack of health insurance
* weight changes > 5 kg in the past 2 months
* pregnancy, breastfeeding
* patients with:

  * severe heart failure
  * impaired hepatic or renal function
  * disturbed coagulation (biopsies will not be taken in those subjects)
  * infection, malabsorption
  * severe hypertension
  * cancer within the last 5 years
  * eating disorders or any other psychiatric condition that would interact with the trial intervention
  * any other endocrine disorder
* changes of smoking habits or diets within the last 3 months prior to study inclusion *other severe chronic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09-12 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Incretine response to different nutritive stimulations | 3 month
  Concentration of GLP-1 after different test meals will be analysed by ELISA before and after weight loss
Incretine response to different nutritive stimulations | 3 month
  Concentration of GIP after different test meals will be analysed by ELISA before and after weight loss
Incretine response to different nutritive stimulations | 3 month
  Concentration of Ghrelin after different test meals will be analysed by ELISA before and after weight loss

SECONDARY OUTCOMES:
Correlation of the GLP-1 responses with the reduction of hunger (questionnaire) after a nutritive stimulation by different nutritional components | 3 month
  GLP-1 (concentration) will be measured by ELISA, hunger feeling will be measured by questionnaire using a visual analog score (from 1 (less) to 10 (more))
correlation of the GIP responses with the reduction of hunger (questionnaire)after a nutritive stimulation by different nutritional components | 3 month
  GIP (concentration) will be measured by ELISA, hunger feeling will be measured by questionnaire using a visual analog score (from 1 (less) to 10 (more))
Correlation of the Ghrelin responses with the reduction of hunger (questionnaire) after a nutritive stimulation by different nutritional components | 3 month
  Ghrelin (concentration) will be measured by ELISA, hunger feeling will be measured by questionnaire using a visual analog score (from 1 (less) to 10 (more))
Correlation of the insulin responses with the reduction of hunger (questionnaire) after a nutritive stimulation by different nutritional components | 3 month
  insulin (concentration) will be measured by ELISA, hunger feeling will be measured by questionnaire using a visual analog score (from 1 (less) to 10 (more))
-differences of substrate utilization depending on the nutritional composition | 3 month
  postprandial thermogenesis will be assessed by indirect caloriemetry
-differences of substrate utilization depending on the nutritional composition | 3 month
  postprandial glucose concentration (physiological parameter) will be assessed in skeletal muscle and adipose tissue by microdialysis
-differences of substrate utilization depending on the nutritional composition | 3 month
  postprandial pyruvate concentration (physiological parameter) will be assessed in skeletal muscle and adipose tissue by microdialysis
-differences of substrate utilization depending on the nutritional composition | 3 month
  postprandial lactate concentration (physiological parameter) will be assessed in skeletal muscle and adipose tissue by microdialysis
-differences of lipolysis depending on the nutritional composition | 3 month
  postprandial glycerol concentration (physiological parameter) will be assessed by microdialysis
-Change of hepatic insulin sensitivity after weight loss | 3 month
  hepatic insulin sensitivity assessed via endogenous glucose production measured in mg/kg/min
-Change of meal induced GLP-1 concentration during weight loss | 3 month
  Concentration of GLP-1 after different test meals will be analysed by ELISA
-Change of meal induced GIP concentration during weight loss | 3 month
  Concentration of GIP after different test meals will be analysed by ELISA
-Change of meal induced Ghrelin concentration during weight loss | 3 month
  Concentration of Ghrelin after different test meals will be analysed by ELISA
-Weight loss mediated changes of meal induced GLP-1 concentration in insulin resistant vs insulin sensitive subjects | 3 month
  Insulin sensitivity assessed via insulin sensitivity index
-Weight loss mediated changes of meal induced GIP concentration in insulin resistant vs insulin sensitive subjects | 3 month
  Insulin sensitivity assessed via insulin sensitivity index
-Weight loss mediated changes of meal induced Ghrelin concentration in insulin resistant vs insulin sensitive subjects | 3 month
  Insulin sensitivity assessed via insulin sensitivity index
Change of fat distribution after weight loss | 3 month
  total fat mass will be assessed
Change of fat distribution after weight loss | 3 month
  visceral fat mass will be assessed
Change of fat distribution after weight loss | 3 month
  hepatic fat mass will be assessed
Change of skeletal muscle mass after weight loss | 3 month
  skeletal muscle mass will be assessed
Prediction of weight regain (weight in kilograms and height in meters will be combined to report BMI in kg/m^2). | 12 months
  Analysis of the predictive impact of hormones like GLP-1, Ghrelin, GIP and insulin in the context of body weight regain. Linear and logistic regression models will be used to identify predictive biomarkers
Prediction of weight regain (weight in kilograms and height in meters will be combined to report BMI in kg/m^2). | 12 months
  Analysis of the predictive impact of hormones like GLP-1, Ghrelin, GIP and insulin in the context of insulin sensitivity. Linear and logistic regression models will be used to identify predictive biomarkers
Prediction of weight regain (weight in kilograms and height in meters will be combined to report BMI in kg/m^2). | 24 months
  Analysis of the predictive impact of hormones like GLP-1, Ghrelin, GIP and insulin in the context of insulin sensitivity. Linear and logistic regression models will be used to identify predictive biomarkers
Prediction of weight regain (weight in kilograms and height in meters will be combined to report BMI in kg/m^2). | 24 months
  Analysis of the predictive impact of hormones like GLP-1, Ghrelin, GIP and insulin in the context of body weight regain. Linear and logistic regression models will be used to identify predictive biomarkers
To analyse the long term course of body weight after 12 month | 12 months
  Measurement of body weight after 12 months
To analyse the long term course of body weight after 24 month | 24 months
  Measurement of body weight after 24 months
To analyse the long term course of body weight after 36 month | 36 months
  Measurement of body weight after 36 months
To analyse the long term course of body weight after 48 month | 48 months
  Measurement of body weight after 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Knut Mai, Prof, Principal Investigator — Charite
Locations (1):
- Charite Campus Mitte, Berlin, Germany

REFERENCES:
- [Derived] Li L, Decker AM, Stobaus N, Beer F, Grittner U, Spranger J, Mai K. Weight loss did not modify macronutrient specific response of hormones and satiety in overweight and obese people without metabolic disease - results from a clinical trial. Clin Nutr. 2022 Apr;41(4):948-957. doi: 10.1016/j.clnu.2022.02.004. Epub 2022 Feb 19. PMID 35303516
- [Derived] Fleischmann R, Decker AM, Kraft A, Mai K, Schmidt S. Mobile electronic versus paper case report forms in clinical trials: a randomized controlled trial. BMC Med Res Methodol. 2017 Dec 1;17(1):153. doi: 10.1186/s12874-017-0429-y. PMID 29191176